CLINICAL TRIAL: NCT07089121
Title: Descartes-08 for Children, Adolescents and Young Adults With Childhood-onset Systemic Lupus Erythematosus, ANCA-associated Vasculitis, Juvenile Myasthenia Gravis, and Juvenile Dermatomyositis
Brief Title: Descartes-08 for Children, Adolescents, and Young Adults With Autoimmune Disorders
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cartesian Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HELIOS-001
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Childhood-onset Systemic Lupus Erythematous; ANCA-Associated Vasculitis (AAV); Juvenile Myasthenia Gravis; Juvenile Dermatomyositis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Dermatomyositis

STUDY DESIGN:
Intervention Model Description: Part 1: establish Maximum tolerated dose Part 2: MTD to be given once weekly for 6 weeks
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Decartes-08 to establish Maximum tolerated dose (Experimental): Intra-patient dose escalation arm with three dose levels over the course of six infusions of cell product.
  Interventions: Drug: Descartes-08
- Part 2: Decartes-08 infusions once weekly for 6 weeks (Experimental): Descartes-08 infusions at the maximum tolerated dose level from Part 1.
  Interventions: Drug: Descartes-08

INTERVENTIONS:
Drug: Descartes-08 — In part 1, three different doses will be administered to 3 participants with either disease indication to establish maximum tolerated dose In part 2, the MTD established in Part-1 will be administered as six once-weekly infusions to up to 10 participants per each of four baskets (cSLE, AAV, JDM and JMG) in an outpatient setting.

SUMMARY:
Safety, tolerability and efficacy of Descarte-08 in children, adolescents and young adults with childhood-onset systemic lupus erythematosus, ANCA-associated vasculitis, juvenile myasthenia gravis, and juvenile dermatomyositis

ELIGIBILITY:
Inclusion Criteria:

* At least age 12
* definitive diagnosis of childhood-onset systemic lupus erythematous, juvenile Myasthenie gravis, juvenile dermatomyositis and AAV
* Signs and symptoms of moderate disease
* History of systemic treatment
* Parent/Guardian/Patient must be able to give written informed consent

Exclusion Criteria:

* Major chronic illness that is not well managed at the time of study entry and in the opinion of the investigator may increase the risk to the patient;
* Abnormal PT/INR or PTT increased > 1.5-fold or patient is on anticoagulation therapy (except in cases of elevated PTT with documented lupus anticoagulant; or in patients who have been on stable doses of anticoagulation therapy for more than 6 months of VTE diagnosis; or in patients on stable doses of anticoagulation therapy for at least 8 weeks of atrial fibrillation diagnosis; these conditions will not be exclusionary unless, in the investigator's opinion, they make participation in the study unsafe);
* ANC < 1000 cells/microliter ;
* Hemoglobin < 8.0 g/dL ;
* Platelets < 50,000/mm3 (NOTE: platelet transfusions are permissible);
* ALT and/or AST with GGT ≥ 3× upper limit of normal
* Creatine Clearance less than 30mL/min /1.73 m2;
* History of primary immunodeficiency, organ, or allogeneic bone marrow transplant;
* Patients must be seronegative for hepatitis B surface antigen;
* Patients must be seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patients must be tested for the presence of viremia by RT-PCR and must be HCV RNA negative;
* History of positive HIV or positive HIV at screening;
* Active tuberculosis or positive QuantiFERON test at screening;
* Any other laboratory abnormality that, in the opinion of the investigator, may jeopardize the subject's ability to participate in the study; 23. Any active significant cardiac or pulmonary disease not related to the primary indication as determined by principal investigator and medical monitor Note: Patients with asthma and COPD controlled with inhaled medications are allowed; 24. Any arterial or venous thromboembolic events in the past 3 months; 25. History of malignancy that required treatment in the past 3 years except for successfully-treated squamous cell and/or basal cell carcinoma of the skin and/or breast or colon cancer that is surgically removed and did not require adjuvant chemotherapy or radiotherapy; 26. Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer); 27. Receipt of a live vaccination within 4 weeks prior to baseline (Day 1) or intent to receive live vaccination during the study (Note: mRNA-based vaccines such as those against SARS-CoV-2 are not considered live; likewise, the Janssen Covid-19 vaccine is not live); 28. History of significant recurrent infections or any active infection that may interfere with the patient's participation in the opinion of the investigator; 29. Any known psychiatric illness that may interfere with the patient's participation in the study in the opinion of the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose in Part 1, type and frequency of treatment related SAE's in Part 2 | Days 22 and 50 for Part1 , Days 22, 50 and Months 3,6,9 and 12 for part 2
  The primary endpoint for Part-1 is the Maximum Tolerated Dose (MTD), defined as the Dose Level at which no more than 20% of the patients treated have shown Dose-Limiting Toxicity (DLT), i.e. at which 3 patients received all 6 weekly infusions without a DLT by Day 50; or 6 patients received 3 weekly infusions with no more than 1 patient having a DLT by Day 50.
  The primary endpoint for Part-2 is the type and frequency of treatment-related SAEs. This will be assessed on Days 22, 50 and Months 3,6,9,12
Maximum Dose Tolerated | Days 2250 for Part 1, Days 11,50, month 3 for part 2 in addition to months, 4,6,9,12
  The primary endpoint for Part-1 is the Maximum Tolerated Dose (MTD), defined as the Dose Level at which no more than 20% of the patients treated have shown Dose-Limiting Toxicity (DLT), i.e. at which 3 patients received all 6 weekly infusions without a DLT by Day 50; or 6 patients received 3 weekly infusions with no more than 1 patient having a DLT by Day 50. The primary endpoint for Part-2 is the type and frequency of treatment-related SAEs.

CONTACTS AND LOCATIONS:
Locations (1):
- H03, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No